CLINICAL TRIAL: NCT01287260
Title: A Multicenter, Double-blind, Parallel-group Comparative Study Between Oral BAYA1040_CR 80 mg and 40 mg for 8 Weeks in Patients With Essential Hypertension for Whom Oral BAYA1040_CR 40 mg is Insufficient
Brief Title: High Dose BAYA1040_Nifedipine: a Dose-comparative Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13176
Record Dates: First submitted 2011-01-30; First posted 2011-02-01 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: BAYA1040_Nifedipine; Nifedipine; Essential hypertension; Japanese Patients; Phase III; 13176
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1 (Experimental)
  Interventions: Drug: Nifedipine (Adalat, BAYA1040)
- Arm 2 (Active Comparator)
  Interventions: Drug: Nifedipine (Adalat, BAYA1040)

INTERVENTIONS:
Drug: Nifedipine (Adalat, BAYA1040) — BAYA1040_Nifedipine 40mg twice daily (BID)
  Arms: Arm1
Drug: Nifedipine (Adalat, BAYA1040) — BAYA1040_Nifedipine 40mg once daily (OD)
  Arms: Arm 2

SUMMARY:
This is a clinical study evaluating the superiority in efficacy and assess safety and tolerability of BAYA1040_Nifedipine 80 mg/day (40 mg twice daily) compared with BAYA1040_Nifedipine 40 mg/day (40 mg once daily) in patients with essential hypertension who are not at target blood pressure by BAYA1040_Nifedipine 40 mg once daily treatment.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* Japanese male or female
* Outpatient with essential hypertension
* Patients whose sitting diastolic blood pressure (DBP) is 90 mmHg or more despite more than 4 weeks of treatment with antihypertensive drug

Exclusion Criteria:

* Sitting diastolic blood pressure (DBP) is 110 mmHg or more or sitting systolic blood pressure (SBP) is 180 mmHg or more
* Patients with secondary hypertension or hypertensive emergency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Efficacy changes measured by sitting diastolic blood pressure (DBP) | Up to 8 weeks

SECONDARY OUTCOMES:
Efficacy changes measured by sitting systolic blood pressure (SBP) | Up to 8 weeks
Achievement rate: Proportion of subjects achieving a target BP based on the Japanese Society of Hypertension (JSH) 2009 guidelines | Up to 8 weeks
Responder rate: Proportion of subjects achieving a target DBP and SBP based on JSH 2009 guidelines or a >10 mmHg reduction of DBP | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Japan (13):
  - Hirosaki, Aomori
  - Kamagaya, Chiba
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Kawasaki, Kanagawa
  - Daitō, Osaka
  - Kishiwada, Osaka
  - Yao, Osaka
  - Tokorozawa, Saitama
  - Shizuoka, Shizuoka
  - Hachiōji, Tokyo
  - Meguro City, Tokyo
  - Minato, Tokyo

REFERENCES:
- [Derived] Shimamoto K, Hasebe N, Ito S, Kario K, Kimura K, Dohi Y, Kawano Y, Rakugi H, Horiuchi M, Imaizumi T, Ohya Y. Nifedipine controlled-release 40 mg b.i.d. in Japanese patients with essential hypertension who responded insufficiently to nifedipine controlled-release 40 mg q.d.: a phase III, randomized, double-blind and parallel-group study. Hypertens Res. 2014 Jan;37(1):69-75. doi: 10.1038/hr.2013.80. Epub 2013 Aug 15. PMID 23945965